CLINICAL TRIAL: NCT04148287
Title: An Open-Label Study to Evaluate the Efficacy and Safety of APX001 in Patients With Candidemia and/or Invasive Candidiasis Caused by Candida Auris
Brief Title: An Open-label Study of APX001 for Treatment of Patients With Candidemia/Invasive Candidiasis Caused by Candida Auris
Acronym: APEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX001-203; C4791011 (Other: Alias Study Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Candidemia; Invasive Candidiases; Candida Infection
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive; Candidiasis

STUDY DESIGN:
Intervention Model Description: Open-label, single arm intervention. All patients will receive APX001. On Days 1-3, APX001 will be administered intravenously. Thereafter, if the patient is able to take oral medication, APX001 tablets will be taken orally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- APX001 (Experimental): APX001 IV or oral for up to 42 days
  Interventions: Drug: APX001

INTERVENTIONS:
Drug: APX001 — Day 1: APX001 1000 mg IV BID over a 3-hour infusion Days 2-3: APX001 600 mg IV QD over a 3-hour infusion Days 4 - 42: APX001 600 mg IV QD over a 3-hour infusion or APX001 800 mg QD oral.
  Other Names: fosmanogepix

SUMMARY:
This is a multicenter, open-label, single arm study to evaluate the efficacy and safety of APX001 for the treatment of candidemia and/or invasive candidiasis caused by C. auris in patients aged 18 years and over with limited antifungal treatment options.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-comparative, single arm study to evaluate the efficacy and safety of APX001 for the treatment of candidemia and/or invasive candidiasis caused by C. auris in patients aged 18 years and over with limited antifungal treatment options. The Study Drug Treatment Period will be up to a maximum of 42 days (inclusive of the loading dose [Study Day 1]). There will be a Follow up Period of 4 weeks (+4 days) after EOST. The total duration of participation in the study is up to approximately 10.5 weeks (inclusive of the Screening Period [168 hours prior to Baseline]).

ELIGIBILITY:
Inclusion Criteria:

* Limited or no treatment options due to resistance, contraindication, intolerance or lack of clinical response to standard of care antifungal therapy, as advocated by the relevant regional/country treatment guidelines
* Established mycological and clinical diagnosis of candidemia and/or invasive candidiasis caused by Candida auris
* Able to have pre-existing intravascular catheters removed and replaced (if necessary)
* Females of childbearing potential with male partners, and males with female partner(s) of childbearing potential, must agree to use 2 forms of highly effective contraception throughout the duration of the study and for 90 days following the last study drug administration. Females of childbearing potential must have a negative urine pregnancy test within 96 hours prior study entry.
* Wiling to participate in the study, willing to give written informed consent, and willing to comply with the study restrictions; where permitted by local regulations, written informed consent from a legal authorized representative (LAR) will be obtained for patients who are unable to give consent

Exclusion Criteria:

* Life expectancy of less than 7 days in the opinion of the Investigator
* Human immunodeficiency virus-infected patients who are receiving antiretroviral therapy that are moderate to strong inducers of CYP3A4, or who have detectable viremia, or who have had an active opportunistic infection within 6 months prior
* Alanine aminotransferase or aspartate aminotransferase greater than or equal to 5 times the upper limit of normal
* Total bilirubin greater than 3 time the upper limit of normal, unless isolated hyperbilirubinemia or due to documented Gilbert's disease
* Pregnant or lactating female patient
* Inappropriate fungal infection source control
* Investigational drug administered within 30 days prior to dosing or five half-lives whichever is longer
* Diagnosis of deep-seated Candida-related infections causing hardware associated septic arthritis, osteomyelitis, endocarditis, myocarditis, hepatosplenic candidiasis, or a central nervous system infection or site of infection that would require antifungal therapy to exceed the maximal duration of study drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (2):
- South Africa (2):
  - Netcare Union Hospital Trauma Surgeons, Alberton, Gauteng
  - Milpark Academic Trauma Centre, Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vazquez JA, Pappas PG, Boffard K, Paruk F, Bien PA, Tawadrous M, Ople E, Wedel P, Oborska I, Hodges MR. Clinical Efficacy and Safety of a Novel Antifungal, Fosmanogepix, in Patients with Candidemia Caused by Candida auris: Results from a Phase 2 Trial. Antimicrob Agents Chemother. 2023 May 17;67(5):e0141922. doi: 10.1128/aac.01419-22. Epub 2023 Apr 6. PMID 37022196

RESULTS

PARTICIPANT FLOW:
Groups:
- APX001 (Fosmanogepix): Participants with candidemia and/or invasive candidiasis caused by Candida auris and with limited antifungal treatment options were administered APX001. On Day 1, participants received APX001 1000 milligrams (mg) as a loading dose over 3 hours by intravenous (IV) infusion twice daily (BID). On Days 2 and 3, participants received APX001 600 mg as maintenance dose over 3 hours by IV infusion once daily (QD). On Day 4 and onwards, maintenance dose was administered as either APX001 600 mg IV infusion QD over 3 hours or APX001 800 mg orally QD. Participants who were clinically stable after 3 days of IV administration and could swallow tablets, could switch from IV to oral dosing from Day 4 and onwards. Maximum treatment duration was of 42 days. Participants were followed up for 4 weeks (+ 4 days) post last dose of study drug.
Period: Overall Study
Arm/Group | APX001 (Fosmanogepix)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- APX001 (Fosmanogepix): Participants with candidemia and/or invasive candidiasis caused by Candida auris and with limited antifungal treatment options were administered APX001. On Day 1, participants received APX001 1000 mg as a loading dose over 3 hours by IV infusion BID. On Days 2 and 3, participants received APX001 600 mg as maintenance dose over 3 hours by IV infusion QD. On Day 4 and onwards, maintenance dose was administered as either APX001 600 mg IV infusion QD over 3 hours or APX001 800 mg orally QD. Participants who were clinically stable after 3 days of IV administration and could swallow tablets, could switch from IV to oral dosing from Day 4 and onwards. Maximum treatment duration was of 42 days. Participants were followed up for 4 weeks (+ 4 days) post last dose of study drug.
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (17.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success at End of Study Treatment (EOST) as Determined by Data Review Committee (DRC)
Description: Treatment success was defined as meeting all of the following criteria:
  1) Two consecutive blood cultures negative for Candida species, and/or for participants with a deep-seated site of infection, at least 1 negative tissue culture or aspirate/fluid culture. For participants with a deep-seated site of infection involving visceral organs from which a tissue culture was not obtainable, resolution of the attributable clinical signs of infection recorded at Baseline, and as applicable, radiological improvement associated with the site of infection. 2) Alive at EOST and 3) No concomitant use of any other systemic antifungal therapies through EOST.
Time Frame: EOST: any day from Day 1 up to maximum of Day 42
Population: The modified intent-to-treat (mITT) population included all participants who received at least 1 dose of study drug and had a confirmed diagnosis of candidemia and/or invasive candidiasis caused by Candida auris within 120 hours (for candidemia) or 168 hours (for invasive candidiasis without candidemia) of study qualification (as determined by the DRC).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Percentage of participants | 88.9 [51.8 to 99.7]

2. Secondary Outcome: Time to First Negative Blood Culture
Description: Time to first negative blood culture was defined as the number of days from date of first dose of study drug to the date of first negative blood culture plus 1. Participants without a negative blood culture at post-baseline visits were censored at the last assessment date. Kaplan-Meier method was used for analysis.
Time Frame: Day 1 up to maximum of Day 42
Population: The mITT population included all participants who received at least 1 dose of study drug and had a confirmed diagnosis of candidemia and/or invasive candidiasis caused by Candida auris within 120 hours (for candidemia) or 168 hours (for invasive candidiasis without candidemia) of study qualification (as determined by the DRC). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 3
Days | 6 [5.0 to 15.0]

3. Secondary Outcome: Percentage of Participants With Mycological Outcomes at EOST and 2 and 4 Weeks After EOST
Description: Mycological outcomes were determined based on eradication and presumed eradication. Eradication was defined as a negative blood (and/or other infection site) culture(s) for Candida species. Presumed eradication (applicable to invasive candidiasis) was defined as clinical resolution of invasive Candida species infection where tissue samples were unavailable. These would be applicable only if there were no concomitant or additional systemic antifungal usage.
Time Frame: EOST: any day from Day 1 up to maximum of Day 42, 2 and 4 weeks after EOST
Population: The mITT population included all participants who received at least 1 dose of study drug and had a confirmed diagnosis of candidemia and/or invasive candidiasis caused by Candida auris within 120 hours (for candidemia) or 168 hours (for invasive candidiasis without candidemia) of study qualification (as determined by the DRC).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Percentage of participants
  EOST | 66.7 [29.9 to 92.5]
  2 Weeks after EOST | 66.7 [29.9 to 92.5]
  4 Weeks after EOST | 66.7 [29.9 to 92.5]

4. Secondary Outcome: Percentage of Participants With Treatment Success at EOST Determined by Investigator
Description: as for outcome 1
Time Frame: EOST: any day from Day 1 up to maximum of Day 42
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Percentage of participants | 88.9 [51.8 to 99.7]

5. Secondary Outcome: Percentage of Participants With Treatment Success at 2 and 4 Weeks After EOST Determined by Investigator and by the DRC
Description: as for outcome 1
Time Frame: 2 and 4 weeks after EOST (where EOST is any day from Day 1 up to maximum of Day 42)
Population: The mITT population included all participants who received at least 1 dose of study drug and had a confirmed diagnosis of candidemia and/or invasive candidiasis caused by Candida auris within 120 hours (for candidemia) or 168 hours (for invasive candidiasis without candidemia) of study qualification (as determined by the DRC). Here, "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure and "number analyzed"= number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 7
Percentage of participants
  2 Weeks after EOST: DRC: number analyzed (Participants) | 6
  2 Weeks after EOST: DRC | 66.7 [29.9 to 92.5]
  4 Weeks after EOST: DRC: number analyzed (Participants) | 6
  4 Weeks after EOST: DRC | 66.7 [29.9 to 92.5]
  2 Weeks after EOST: Investigator | 77.8 [40.0 to 97.2]
  4 Weeks after EOST: Investigator | 77.8 [40.0 to 97.2]

6. Secondary Outcome: All-Cause Mortality Through Study Day 30
Description: Percentage of participants who died through study Day 30 is reported in this outcome measure.
Time Frame: Day 1 through Day 30
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Percentage of participants | 11.1

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between first dose of study drug and up to Week 4 (+4 days) post last dose of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to maximum of 32 days of follow up post last dose of study drug, where maximum treatment duration was 42 days (maximum up to 74 days)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix)
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 32 days of follow up post last dose of study drug, where maximum treatment duration was 42 days (maximum up to 74 days)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | APX001 (Fosmanogepix)
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APX001 (Fosmanogepix) (N=9)
Cardiac arrest (Cardiac disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Pneumonia (Infections and infestations) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APX001 (Fosmanogepix) (N=9)
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Generalised oedema (General disorders) | 1
Hypothermia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04148287/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04148287/SAP_003.pdf